CLINICAL TRIAL: NCT01394510
Title: Effect of Anti-oxidants on Beta-cell Function in Humans
Brief Title: Effect of the Anti-oxidant N-acetylcysteine on Beta-cell Function in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Utzschneider, Kristina, M.D. (Individual)
Collaborators: VA Puget Sound Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kristina Utzschneider, MD, Associate Professor of Medicine, Utzschneider, Kristina, M.D.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NACStudy001
Record Dates: First submitted 2011-07-12; First posted 2011-07-14 (Estimated); Results first posted 2016-06-17 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-05

CONDITIONS: Type 2 Diabetes; Oxidative Stress
Keywords: insulin secretion; beta-cell function; oxidative stress; type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- N-acetylcysteine dose study (Experimental): Subjects will take N-acetylcysteine (NAC) 600 mg twice daily for 2 weeks, then 1200 mg twice daily for an additional 2 weeks. Study procedures will be performed at baseline, after 2 weeks and after 4 weeks.
  Interventions: Drug: N-acetylcysteine

INTERVENTIONS:
Drug: N-acetylcysteine — 600 mg N-acetylcysteine (NAC) twice daily by mouth for 2 weeks followed by 1200 mg NAC twice daily by mouth for 2 additional weeks.
  Other Names: NAC

SUMMARY:
Insulin is secreted by cells in the pancreas called beta-cells. Beta-cell dysfunction is a critical feature of type 2 diabetes (T2DM). High glucose levels can exacerbate beta-cell dysfunction with oxidative stress proposed as a major mediator of this "glucotoxic" effect. High glucose levels have also been shown to contribute to vascular dysfunction and inflammation and these adverse responses decreased with the use of antioxidants. The hypothesis is that antioxidants improve beta-cell function in individuals with elevated glucose levels by decreasing oxidative stress. In this study the investigators will specifically test whether the antioxidant N-acetylcysteine (NAC) can improve beta-cell function in individuals with type 2 diabetes by decreasing oxidative stress.

This study will be a dose finding study to determine the tolerability of 600 mg versus 1200 mg twice a day of NAC and the effects on beta-cell function, glucose tolerance and oxidative stress markers in persons with type 2 diabetes.

DETAILED DESCRIPTION:
Beta-cell dysfunction is a critical feature of type 2 diabetes (T2DM). High glucose levels can exacerbate beta-cell dysfunction with oxidative stress proposed as a major mediator of this "glucotoxic" effect. High glucose levels have also been shown to contribute to vascular dysfunction and inflammation and these adverse responses decreased with the use of antioxidants. The hypothesis is that antioxidants improve beta-cell function in individuals with elevated glucose levels by decreasing oxidative stress. In this study the investigators will specifically test whether the antioxidant N-acetylcysteine (NAC) can improve beta-cell function in individuals with type 2 diabetes by decreasing oxidative stress.

This initial study will be a dose finding study to determine the tolerability of 600 mg versus 1200 mg twice a day of NAC and the effects of NAC treatment on beta-cell function, glucose tolerance and oxidative stress markers in persons with type 2 diabetes. Study procedures will include a fasting urine sample and performance of a 2 hour 75 gram oral glucose tolerance test at baseline, after 2 weeks on 600 mg twice daily NAC and again after 2 more weeks on 1200 mg NAC twice a day.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes

Exclusion Criteria:

* Pregnant or lactating females
* Uncontrolled diabetes mellitus with severe hyperglycemia (hemoglobin A1C ≥ 9%)
* Patients with diabetes mellitus who are taking insulin or glucose-lowering agents other than metformin
* Chronic oral or parenteral corticosteroid treatment (>7 consecutive days of treatment) within 8 weeks prior to screening
* Use of human immunodeficiency virus (HIV) protease inhibitors or niacin
* Chronic inflammatory diseases or use of anti-inflammatory drugs.
* Thyroid abnormalities (thyroid-stimulating hormone [TSH] <0.5 or >5 µU/ml)
* Creatinine >1.5 in men and >1.3 mg/dl in women
* History of dysphagia, gastroparesis, gastric ulcer, malabsorption, swallowing disorders or intestinal motility disorder
* Gastroesophageal reflux disease (heartburn) requiring treatment.
* Active cancer
* Clinical hepatic disease or alanine aminotransferase (ALT) greater than ≥ 1.5 times upper limit of normal within 60 days preceding the first dose of the study drug
* Weight loss of >5% body weight within the last 6 months, or starting an intensive exercise program within 4 weeks of study initiation
* Smoke or use tobacco
* Excessive alcohol consumption (>2 drinks a day)
* Use of any investigational drug in the last 30 days
* Anemia (hematocrit <33%), donation of one unit (500 ml) or more of blood, significant blood loss equaling at least one unit of blood within the past 2 weeks or a blood transfusion within 8 weeks prior to screening
* Employment by the research center

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-06; Primary Completion 2014-09 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Utzschneider, MD, Principal Investigator — VA Puget Sound Health Care System
Locations (1):
- VA Puget Sound Health Care System, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
The study sample size is very small. The data will be made available upon request.

REFERENCES:
- [Result] Szkudlinska MA, von Frankenberg AD, Utzschneider KM. The antioxidant N-Acetylcysteine does not improve glucose tolerance or beta-cell function in type 2 diabetes. J Diabetes Complications. 2016 May-Jun;30(4):618-22. doi: 10.1016/j.jdiacomp.2016.02.003. Epub 2016 Feb 5. PMID 26922582

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | N-acetylcysteine Dose Study
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients with type 2 diabetes either on metformin alone or treated with diet and lifestyle only.
Arm/Group | N-acetylcysteine Dose Study
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 6
body mass index [Mean (Standard Deviation); unit: kg/m2] — Body mass index
  kg/m2 | 37.3 (10.1)
HbA1c [Mean (Standard Deviation); unit: %] | 6.17 (2.05)
metformin [Number; unit: participants] — number of patients taking metformin
  participants | 6

OUTCOME MEASURES:

1. Primary Outcome: Fasting Urine F2 Alpha Isoprostane Levels
Description: Change in fasting urine isoprostane levels at 4 weeks vs baseline as a marker of oxidative stress
Time Frame: 4 weeks
Population: Change in urine F2 alpha isoprostanes/mg urine creatinine. Urine isoprostanes were only measured in a subset of participants due to lack of effect of the intervention on glucose tolerance.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | N-acetylcysteine Dose Study
Number analyzed (Participants) | 9
ng/ml | -0.089 (1.28)

2. Secondary Outcome: Area Under the Curve for Glucose (AUCg)
Description: Change in AUCg from 0-120 minutes during the oral glucose tolerance test at 4 weeks compared to baseline
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: mg/dl x 120 minutes
Arm/Group | N-acetylcysteine Dose Study
Number analyzed (Participants) | 13
mg/dl x 120 minutes | -1011 (10922)

3. Secondary Outcome: Oral Disposition Index
Description: The change in the oral disposition index defined was the change in the early insulin response divided by the change in glucose from 0-30 minutes during the oral glucose tolerance test divided by fasting insulin.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | N-acetylcysteine Dose Study
Number analyzed (Participants) | 12
mg/dl | -0.08 (0.18)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | N-acetylcysteine Dose Study
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No